CLINICAL TRIAL: NCT05137080
Title: Dexamethasone and Functional Outcome After Total Knee Arthroplasty: A 2 Year Follow up of the DEX-2-TKA-trial
Brief Title: Dexamethasone and Functional Outcome After TKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Slagelse Hospital (Other)
Responsible Party: Principal Investigator, Asger Krog Moelgaard, MD, Ph.D.-student, Slagelse Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-RCAI-ASMAN-st02; SJ-944 (Other: Regional Ethics Committee); REG-108-2021 (Other: List of ongoing research in Region Zealand (on behalf of the Danish Data Protection Agency))
Record Dates: First submitted 2021-11-16; First posted 2021-11-30 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Chronic Knee Pain; Dexamethasone; Total Knee Arthroplasty
MeSH Terms: interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment A (Active Comparator): 24mg dexamethasone i.v. perioperatively and 24mg dexamethasone i.v. on the first postoperative day
  Interventions: Drug: Dexamethasone
- Treatment B (Active Comparator): 24mg dexamethasone i.v. perioperatively and placebo (isotonic saline) i.v. on the first postoperative day
  Interventions: Drug: Dexamethasone; Drug: Isotonic saline
- Treatment C (Placebo Comparator): Placebo (isotonic saline) i.v. perioperatively and placebo (isotonic saline) i.v. on the first postoperative day
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: Dexamethasone — 24mg dexamethasone
  Arms: Treatment A; Treatment B
Drug: Isotonic saline — Isotonic saline
  Arms: Treatment B; Treatment C

SUMMARY:
Patients previously included in the DEX-2-TKA-trial (ethics committee ID SJ-695; ClinicalTrials.gov: NCT03506789) at Næstved Hospital will be invited for a follow up study consisting of questionnaires and a visit with a physical therapist. The study includes the following validated questionnaires: EQ-5D-5L, Oxford Knee Score and PainDetect, and information on height, weight, daily pain-medication and co-morbidities. With the physical therapist, the patient will perform the following functional tests: knee range of motion, timed-up-to-go, 30 second chair stand test, 40m fast paced walk test, stair climb test and a measure of the thigh force.

ELIGIBILITY:
Inclusion Criteria:

* participation in the DEX-2-TKA-trial at Næstved Hospital in accordance with protocol
* Signed, informed consent for participation

Exclusion Criteria:

* Lack of signed, informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Average pain during functional performance exercises | 2-3 years after total knee arthroplasty
  Average of maximal pain experienced during the functional performance exercises measured as a VAS 0-100mm with comparisons between treatment allocation group. The average will be calculated based on measurements after each functional performance exercise (TUG, 30CST, 40FPW and SCT).

SECONDARY OUTCOMES:
EQ-5D-5L | 2-3 years after total knee arthroplasty
  Difference in performance between treatment allocation groups on the EQ-5D-5L questionnaire at follow-up. EQ-5D-5L is comprised of five health dimensions (mobility, self-care, usual activities, pain/discomfort) which the patient must rate on a 1-5 dimension going from no problems to perform the activity to being unable to perform the activity. In addition, the patient will rate his/her health on a 0-100 scale, where 0 being worst imaginable health and 100 being best imaginable health.
Oxford Knee Score | 2-3 years after total knee arthroplasty
  Difference in performance between allocation groups on the Oxford Knee Score questionnaire at follow-up. Oxford Knee Score is a questionnaire comprised of 12 questions regarding pnee pain and function. Each question can be answered on a 1 (best) to 5 (worst) score and thus a overall scores can be calculated by summing op all the scores. Best outcome would hence be a score of 12, while worst possible outcome is a score of 60.
PainDetect | 2-3 years after total knee arthroplasty
  Difference in performance between allocation groups on the PainDetect questionnaire at follow-up. The PainDetect questionnaire is comprised of 11 questions regarding strengt and character of any experienced pain. The patients answers can then be calculated into a total score of 0-38 and further grouped into likelihood of a neuropathic component of the patients chronic pain. If 0-12 there is <15% likelihood that the patient experiences neuropathic pain, while >18 estimates a likelihhed >90% for a neuropathic component. 13-18 points is a greyzone in between where a neuropathic component of the experienced pain cannot either be ruled in or out.
Use of opioids | 2-3 years after total knee arthroplasty
  Difference in daily use of opioids between allocation groups at follow-up. Daily use will be calculated into equivalents of mg morphine per day.
Range of Motion | 2-3 years after total knee arthroplasty
  Difference in performance between allocation groups on the Range of Motion exercise at follow-up. Range of motion is measured in degrees from fully extended to full flexion of the knee
Timed-Up-To-Go (TUG) | 2-3 years after total knee arthroplasty
  Difference in performance between allocation groups on the timed-up-to-go-test exercise at follow-up assessed as time in seconds it takes to
  * Stand up from the chair
  * Walk to a line on the floor 3 meters away
  * Turn
  * Walk back to the chair
  * Sit down again. The time will be measured from "Go" to the participant is sitting again.
30 second chair stand test (30CST) | 2-3 years after total knee arthroplasty
  Difference in performance between allocation groups on the 30 second chair-stand-test exercise at follow-up assessed as number of repetitions performed during 30 seconds. one repetition is counted as
  * sitting on a chair with the arms crossed across the chest
  * stand fully up
  * sit down again
40 meter fast paced walk test (40FPW) | 2-3 years after total knee arthroplasty
  Difference in performance between allocation groups on the 40 meter fast paced walk test exercise at follow-up assessed as walk speed in meters pr. second. The exercised is performed by the patient walkning as highest possible speed between to lines on the floor 10 meters apart from each other. A timer is started eache time the patient crossess the line and paused, when the patient is at the other end. After 4 walks between the lines the 40 meters is divided by the total time in seconds and expressed as meters pr. second
Stair Climb Test (SCT) | 2-3 years after total knee arthroplasty
  Difference in performance between allocation groups on the stair climb test exercise at follow-up assessed as time in seconds it takes to walk 9 steps up and 9 steps down a flight of stairs.
Thigh Force | 2-3 years after total knee arthroplasty
  Difference in thigh force between allocation groups at follow-up assessed during flexion and extension. Force will be measured with an EASYFORCE-apparatus and expressed as newton.

CONTACTS AND LOCATIONS:
Overall Officials: Asger K Mølgaard, MD, Principal Investigator — Research Center for Anaesthesiology and Intensive Care Medicine, Department of Anaesthesiology, Næstved, Slagelse and Ringsted Hospitals; Daniel Hägi-Pedersen, MD, Ph.D., Study Chair — Research Center for Anaesthesiology and Intensive Care Medicine, Department of Anaesthesiology, Næstved, Slagelse and Ringsted Hospitals; Kasper S Gasbjerg, MD, Study Chair — Research Center for Anaesthesiology and Intensive Care Medicine, Department of Anaesthesiology, Næstved, Slagelse and Ringsted Hospitals; Ole Mathiesen, MD, PhD, Assoc Prof, Study Chair — Centre for Anaesthesiological Research, Department of Anaesthesiology, Zealand University Hospital; Søren T Skou, PhD, Assoc Prof, Study Chair — PROgrez, Department of physical therapy and Occupational Therapy, Næstved, Slagelse and Ringsted Hospitals
Locations (2):
- Denmark (2):
  - Næstved, Slagelse og Ringsted Hospitals, Næstved
  - Næstved, Slagelse and Ringsted Hospitals, Slagelse

IPD SHARING:
Plan to Share IPD: Undecided
If data are to be published, they will be anonymised according to ICIMEs (International Committee of Medical Journal Editors) guidelines

REFERENCES:
- [Derived] Molgaard AK, Gasbjerg KS, Skou ST, Mathiesen O, Hagi-Pedersen D. Chronic Pain and Functional Outcome 3 years After Total Knee Arthroplasty and Perioperative Dexamethasone: A Follow-Up of the Randomized, Clinical DEX-2-TKA Trial. J Arthroplasty. 2023 Dec;38(12):2592-2598.e2. doi: 10.1016/j.arth.2023.05.060. Epub 2023 Jun 5. PMID 37286048